CLINICAL TRIAL: NCT00220428
Title: The Effect of T-Cell Vaccination in Multiple Sclerosis - Phase I/II Safety and Efficacy Trial
Brief Title: T-Cell Vaccination in Multiple Sclerosis (MS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: SHEBA-98-1754-AA-CTIL
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Multiple Sclerosis
Keywords: T cell
MeSH Terms: conditions — Multiple Sclerosis

INTERVENTIONS:
Biological: T-Cell Vaccination

SUMMARY:
The purpose of this study is to evaluate the safety of T-cell vaccination in MS patients.

DETAILED DESCRIPTION:
Immunization of MS patients with irradiated autologous encephalitogenic myelin peptides (EMP) specific T-cell lines or clones.

Clinical immunologic and neuroradiologic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS (post criteria)
* Relapsing remitting or primary progressive clinical course. At least one relapse in the last two years.
* Disease duration > 1 year
* Expanded Disability Status Scale (EDSS) between 0-6
* Brain magnetic resonance imaging (MRI) compatible with MS
* Not involved in any other clinical trials
* No other systemic disease

Exclusion Criteria:

* Does not comply with the above

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 1998-07; Study Completion 2007-12

PRIMARY OUTCOMES:
safety assessment of T-cell vaccination in nonresponding MS patients

CONTACTS AND LOCATIONS:
Overall Officials: Anat Achiron, MD PhD, Principal Investigator — Sackler School of Medicine
Locations (1):
- Multiple Sclerosis Center, Ramat Gan, Israel